CLINICAL TRIAL: NCT01953120
Title: Mechanisms of Belatacept (Nulojix) Effect on Alloimmunity and Antiviral Response After Kidney Transplantation - (BMS Study# IM 103-309)
Brief Title: Mechanisms of Belatacept Effect on Alloimmunity and Antiviral Response After Kidney Transplantation (BMS IM 103-309)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Suphamai Bunnapradist, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-000270
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Renal Transplant Rejection
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belatacept (Experimental): Survival and rejection in patients switched to belatacept.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Subjects will receive intravenous belatacept at 5mg/kg every other week starting from day 1 and continuing with weeks 2, 4, 6, and 8, and then monthly at months 3, 4, 5, and 6. At month 6 patients may elect to continue for an additional six-month period of belatacept administration.
  Other Names: Nulojix

SUMMARY:
This research evaluates the effectiveness of a new drug called belatacept (Nulojix) for the prevention of acute rejection and preservation of kidney function in transplant patients. Belatacept was approved in 2011 by the United States Food and Drug Administration (FDA) and is being marketed as Nulojix. The pharmaceutical company sponsoring this study is Bristol-Myers Squibb.

Belatacept is a prescription medicine used in adults to prevent transplant rejection in people who have received a kidney transplant. Transplant rejection happens when the body's immune system senses that the new transplanted kidney is different or foreign, and attacks it. Belatacept is used with corticosteroids and certain other medicines to help prevent rejection of your new kidney.

The purpose of the research is to understand whether the new drug, belatacept, is better than other anti-rejection drugs, such as cyclosporine and tacrolimus that are typically used in the treatment against kidney rejection in transplant patients.

DETAILED DESCRIPTION:
Research Hypothesis: Switching to a belatacept-based immunosuppression regimen after kidney transplant will have a significant impact on antibody and T cell-mediated immune response as compared with control patients as measured in peripheral blood at 6 months after belatacept switch and comparable safety and efficacy as compared with calcineurin inhibitor (CNI) based regimens.

Primary Objective: To analyze the effect of switching from CNI to belatacept in patients with evidence of CNI toxicity on the development and maintenance of immune memory in response to both alloantigen and viral antigens commonly encountered after transplant, and to assess the safety and efficacy of conversion to belatacept as maintenance immunosuppression in combination with prednisone and mycophenolate mofetil.

Study Design: Open label, single center clinical trial. Patients with evidence of CNI toxicity will be eligible for switch to belatacept-based regimen within the first three months after transplant. All enrolled subjects will also receive concomitant maintenance immunosuppression with mycophenolate mofetil and corticosteroids.

Duration of Study: 6 months, with option to extend to 12 months of belatacept treatment Number of Subjects: 20 Study Population: Kidney transplant recipients within the first three months of their first transplant with evidence of CNI toxicity.

Test Product, Dose and Mode of Administration, Duration of Treatment: Study patients will receive intravenous belatacept at 5mg/kg every two weeks at day 1 and weeks 2, 4, 6, and 8, and then monthly at months 3, 4, and 5. At month 6 patients may elect to continue for an additional six month period of belatacept administration. Peripheral blood mononuclear cells (PBMCs) and sera for antibody testing will be collected at time of study entry and at 4, 8, 12, and 24 weeks after belatacept start, frozen and banked at our center, and analyzed in batch fashion for development of humoral and cell mediated immunity. Patients who elect to receive an additional 6 months of belatacept treatment will undergo additional immunologic analysis at 1 year after study entry.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing to provide signed written informed consent Target Population
2. The subject is a first-time recipient of a living or deceased donor kidney transplant
3. Evidence of calcineurin inhibitor side effects during the first 3 months after transplant as defined as

1. Neurologic toxicity, defined as tremor, altered mental status, or seizure 2. Renal toxicity, defined as glomerular filtration rate (GFR) <60 3. Metabolic toxicity, defined as a new requirement for medication to control hyperglycemia 4. Hematologic toxicity, defined as development of thrombotic microangiopathy Age and Gender 4) Men and women, ages 18 and older, inclusive 5) Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study in such a manner that the risk of pregnancy is minimized. Refer to the protocol for details regarding description and handling of WOCBP subjects.

WOCBP must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin (HCG)) within 72 hours prior to the start of study medication then every 3 months during the period of study participation.

6) Men must use an adequate method of contraception throughout the study, and for up to 8 weeks after the last infusion, so that the risk of pregnancy to their partners is minimized.

7) Mycophenolate mofetil (MMF) must be dosed at 500 mg by mouth twice daily or greater at the time of study entry 8) Prednisone must be dosed at >=10 mg by mouth daily for patients less than 6 weeks post-transplantation, and at >=5mg by mouth daily for patients greater than 6 weeks post-transplantation at the time of study entry.

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last infusion.
2. Women who are pregnant or breastfeeding
3. Women with a positive pregnancy test on enrollment or prior to study drug administration
4. Males unwilling or unable to use an adequate method of contraception for the entire study period and for up to 8 weeks after the last infusion of study medication Immunologic status
5. Subjects with panel reactive antibody (PRA) ≥ 30% at time of transplant
6. Subjects with zero human leukocyte antigen (HLA) mismatched donors (either from related or unrelated donor)
7. Subjects with any prior solid organ transplant (including kidney)
8. Subjects receiving a concurrent solid organ (heart, liver, pancreas) or cell (islet, bone marrow, stem cell) transplant
9. Subjects with a history of biopsy-proven acute rejection post-transplant (humoral or cellular) in the first three months post transplantation Infection related risks
10. Subjects who are hepatitis C antibody-positive or polymerase chain reaction (PCR)-positive for hepatitis C
11. Subjects who are hepatitis B surface antigen-positive or PCR-positive for hepatitis B
12. Subjects with known human immunodeficiency virus (HIV) infection
13. Subjects with active tuberculosis (TB) requiring treatment within the previous 3 years or any subject who previously required triple (or more) combination therapy for TB.
14. Subjects who are Epstein-Barr virus (EBV) antibody negative and have received grafts from EBV antibody positive donors.

    Prohibited Therapies and/or Medications
15. Subjects who have used any investigational drug within 30 days prior to the Day 1 visit
16. Subjects previously treated with belatacept
17. Use of mammilian target of rapamycin (mTOR) inhibitors at any time after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2021-04 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suphamai Bunnapradist, M.D., Principal Investigator — UCLA Kidney Transplant Research
Locations (1):
- UCLA Kidney Transplant Research, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schaenman J, Rossetti M, Pickering H, Sunga G, Wilhalme H, Elashoff D, Zhang Q, Hickey M, Reddy U, Danovitch G, Reed EF, Bunnapradist S. Preservation of Antiviral Immunologic Efficacy Without Alloimmunity After Switch to Belatacept in Calcineurin Inhibitor-Intolerant Patients. Kidney Int Rep. 2022 Oct 20;8(1):126-140. doi: 10.1016/j.ekir.2022.10.015. eCollection 2023 Jan. PMID 36644348

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Belatacept
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Belatacept
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 8
Induction, Anti-thymocyte globulin (ATG) [Count of Participants; unit: Participants] | 6
Deceased Donor [Count of Participants; unit: Participants] | 8
Cytomegalovirus (CMV) Seropositive [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Antibody and T Cell-mediated Immune Response
Description: To analyze the effect of switching from CNI to belatacept in patients with evidence of CNI toxicity on the development and maintenance of immune memory in response to both alloantigen and viral antigens commonly encountered after transplant, and to assess the safety and efficacy of conversion to belatacept as maintenance immunosuppression in combination with prednisone and mycophenolate mofetil.
Time Frame: Month 6
Population: Clinical outcomes measured included CMV viremia, PTLD, development of donor specific antibodies, acute rejection, and death. Laboratory based measurements included immune phenotype, alloimmune response as measured by intracellular cytokine stimulation (ICS), and antiviral immune response to CMV and EBV as measured by ICS.
Measure: Number; unit: participants
Arm/Group | Belatacept
Number analyzed (Participants) | 19
participants
  CMV Viremia | 17
  PTLD | 0
  Development of Donor Specific Antibodies | 0
  Acute Rejection | 1
  Death | 0

2. Secondary Outcome: Post-transplant de Novo Donor Specific Antibody (DSA)
Description: Incidence of de novo DSA detected at one or more time points during the period of study
Time Frame: Months 1, 3, and 12 if applicable as the secondary measures continue belatacept treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept
Number analyzed (Participants) | 19
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected over 12 months.
Description: Serious Adverse Events were defined per protocol as: results in death.
Arm/Group | Belatacept
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT01953120/Prot_SAP_000.pdf